CLINICAL TRIAL: NCT07116668
Title: SafeHeal Colovac Anastomosis Protection Device Evaluation (SAFE-3CV) Pivotal Study: A Study to Evaluate Safety and Effectiveness of the Colovac Anastomosis Protection Device
Brief Title: SafeHeal Colovac Anastomosis Protection Device Evaluation Pivotal Study
Acronym: SAFE-3CV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: SafeHeal Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-3CV
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Stoma - Ileostomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The SafeHeal Colovac Anastomosis Protection Device Evaluation (SAFE-3CV) Pivotal Study is a prospective, non-randomized, sequential, IDE multicenter trial enrolling patients who are implanted with the investigational device, the Colovac Anastomosis Protection Device (next generation). These patients will be compared to a control group, the standard of care (diverting ostomy) and analyzed using a propensity subclassification approach with pre-specified covariates. The control data were collected as part of the SH-SOC23 study, a prospective, non-randomized, multicenter study sponsored by SafeHeal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Colovac arm (Experimental): Subjects treated with the Colovac Device following low anterior resection of the colon will be enrolled in the investigational cohort.
  Interventions: Device: Colovac Anastomosis Protection Device placement following low anterior resection of colon cancer

INTERVENTIONS:
Device: Colovac Anastomosis Protection Device placement following low anterior resection of colon cancer — Subjects in the Investigational cohort (SAFE-3CV) will undergo an LAR procedure followed by Colovac placement. Colovac retrieval will then occur at ~10 days post LAR procedure.

SUMMARY:
Colorectal cancer is the third most common malignancy worldwide and the second most common in the US. It is the second leading cause of cancer death worldwide, with 1.8 million new cases and 862,000 deaths per year. The majority of patients receive surgical treatment. Colorectal surgery is associated with a high risk of morbidity and mortality in comparison to other general surgery subspecialties. This study aims to further assess the safety and effectiveness of the Colovac Anastomosis Protection Device, a temporary intraluminal bypass device, on a larger scale.

DETAILED DESCRIPTION:
The Colovac Anastomosis Protection Device is intended for use in patients requiring low anterior rectal anastomoses to limit stoma creation to only those patients requiring more time for anastomosis healing when the device is removed, allowing patients with a healed anastomosis to avoid stoma creation. To reduce the risk of life-threatening complications, Colovac provides an alternative to stoma creation which prevents stoma related risks, including permanent stoma.

ELIGIBILITY:
Inclusion Criteria:

A subject meeting all of the following criteria will be considered for participation in the study:

1. Adult patients (22 years of age or older)
2. Eligible to undergo open or minimally invasive sphincter-sparing low anterior resection with planned diverting loop ileostomy for malignancy.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
4. Willingness to comply with protocol-specific treatment and study visits and to sign a written Informed Consent Form

Exclusion Criteria:

* Preoperative:

  1. Active colitis
  2. Known allergy to nickel or other components of the Colovac system
  3. Pregnant or nursing female subject
  4. Concomitant major surgical procedure in combination with Colorectal resection (i.e., hepatectomy)
  5. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation, impair the ability of the participant to undergo protocol-described procedures or interfere with the interpretation of study results including, but not limited to:

     1. Stage IV colorectal cancer unless curative intent R0 resection is planned AND there is no associated peritoneal disease
     2. Immunodeficiency (CD4+ count < 500 CU MM)
     3. Systemic and ongoing steroid therapy within the past 6 months
     4. Systemic infection at the time of surgery or requiring systemic antimicrobial therapy up to 1 week before surgery
     5. Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
     6. Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel, or carcinomatosis
     7. Fecal incontinence, involvement of sphincter by the neoplastic disease or evidence of extensive local disease in the pelvis seen on pre-operative imaging
     8. Severe malnutrition defined as 10% weight loss within 3 months prior to enrollment.
  6. The subject is currently participating in another investigational drug or device study that may confound the results of SAFE-3CV. Prior approval from SafeHeal Medical Monitor must be obtained prior to enrollment in SAFE-3CV.

     Intraoperatively:
  7. Occurrence of any of the following during the colorectal surgery:

     1. Blood loss (>750 cc)
     2. Blood transfusion
     3. Any new sign of bowel ischemia
     4. Positive air leak test
     5. Inadequate bowel preparation
     6. Anastomosis location greater than 10 cm from the anal verge
     7. Any other surgical complications or intra-operative risks that may place the patient at greater risk from study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Performance: Clinically meaningful ostomy avoidance rate at Day 10 | at 10 day visit
  The primary performance endpoint assessed for Colovac subjects at the Day 10 visit is a clinically meaningful ostomy avoidance rate that supports a favorable benefit risk when considering the primary safety endpoint.
Safety: Cumulative rate of Major Complications | 9 months
  The primary safety endpoint is the cumulative rate of subjects with major complications through 9 months.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (13):
  - Kaiser Permanente, Los Angeles, California
  - Keck Medicine of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Mount Sinai Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Novant Health, Winston-Salem, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
- Belgium (2):
  - UZA, Edegem, Antwerp
  - UZ Leuven, Leuven, Flemish Brabant
- France (3):
  - Chu du Rouen, Rouen, Normandy
  - Bordeaux Colorectal Institute, Bourdeaux, Nouvelle-Aquitaine
  - Hopital Saint-Antoine, Paris, Île-de-France Region
- Humanitas Research Hospital, Rozzano, Lombardi, Italy